CLINICAL TRIAL: NCT03474471
Title: A Prospective Randomized Controlled Trial on the Systemic Effects of Bronchoscopic Lung Volume Reduction in Patients With Severe Emphysema.
Brief Title: A Trial on the Effects of Bronchoscopic Lung Volume Reduction in Severe Emphysema.
Acronym: SOLVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Maastricht University Medical Center (Other); Center of Expertise for Chronic Organ Failure (Other)
Responsible Party: Principal Investigator, Dirk-Jan Slebos, dr. D.J. Slebos, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOLVE
Record Dates: First submitted 2018-03-09; First posted 2018-03-22 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Emphysema
MeSH Terms: conditions — Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1:PR-EBV treatment (Experimental): Follow a Pulmonary rehabilitation program PRIOR to the EBV treatment
  Interventions: Behavioral: Pulmonary rehabilitation; Device: EBV treatment
- Group 2: EBV treatment-PR (Experimental): Follow a Pulmonary rehabilitation program AFTER the EBV treatment
  Interventions: Behavioral: Pulmonary rehabilitation; Device: EBV treatment
- Group 3: EBV treatment (Active Comparator): Only EBV treatment
  Interventions: Device: EBV treatment

INTERVENTIONS:
Behavioral: Pulmonary rehabilitation — Following a PR program
  Arms: Group 1:PR-EBV treatment; Group 2: EBV treatment-PR
Device: EBV treatment — Bronchoscopic lung volume reduction using endobronchial valves (EBV)

SUMMARY:
Rationale: The published clinical trials investigating the bronchoscopic lung volume reduction, showing important patient-related improvements in efficacy, led to the acknowledgement of the treatment in the GOLD-COPD2017 guidelines. Interaction with pulmonary rehabilitation, impact on patient-reported outcomes, physical activity, and extrapulmonary consequences are all topics to gain more insight in. This importantly, to further develop and optimize this innovative and personalized therapy.

Objective: To study in detail the impact and optimal timing of pulmonary rehabilitation (PR) on exercise physiology and patient-reported outcomes and the impact of the bronchoscopic lung volume reduction treatment using endobronchial valves (EBV) on cardiopulmonary function, metabolism and changes in body composition.

Study design: This study is a randomized controlled trial with 3 study-arms. Group 1 will first follow a PR program and afterwards undergo the EBV treatment. Group 2 will first undergo the EBV treatment and approximately 8 weeks later will follow a PR program. Group 3 will only undergo the EBV treatment (and can choose to follow a PR program after completing the 6 month FU visit).

Study population: The study population exist of patients with severe emphysema who undergo a bronchoscopic lung volume reduction treatment using one-way valves.

Intervention: Most patients will undergo a bronchoscopic lung volume reduction treatment using endobronchial valves and a pulmonary rehabilitation program. One group of patient will under a bronchoscopic lung volume reduction treatment using endobronchial valves and can choose whether they also want to follow a pulmonary rehabilitation program afterwards.

Main study parameters: The main study parameter is the difference in change in endurance time measured by an endurance cycle test between the EBV treatment group and the bronchoscopic lung volume reduction + rehabilitation group (EBV+PR).

DETAILED DESCRIPTION:
Rationale: The published clinical trials investigating the bronchoscopic lung volume reduction, showing important patient-related improvements in efficacy, led to the acknowledgement of the treatment in the GOLD-COPD2017 guidelines. Interaction with pulmonary rehabilitation, impact on patient-reported outcomes, physical activity, and extrapulmonary consequences are all topics to gain more insight in. This importantly, to further develop and optimize this innovative and personalized therapy.

Objective: To study in detail the impact and optimal timing of pulmonary rehabilitation (PR) on exercise physiology and patient-reported outcomes and the impact of the bronchoscopic lung volume reduction treatment using endobronchial valves (EBV) on cardiopulmonary function, metabolism and changes in body composition.

Study design: This study is a randomized controlled trial with 3 study-arms. Group 1 will first follow a PR program and afterwards undergo the EBV treatment. Group 2 will first undergo the EBV treatment and approximately 8 weeks later will follow a PR program. Group 3 will only undergo the EBV treatment (and can choose to follow a PR program after completing the 6 month FU visit).

Study population: The study population exist of patients with severe emphysema who undergo a bronchoscopic lung volume reduction treatment using one-way valves.

Intervention: Most patients will undergo a bronchoscopic lung volume reduction treatment using endobronchial valves and a pulmonary rehabilitation program. One group of patient will under a bronchoscopic lung volume reduction treatment using endobronchial valves and can choose whether they also want to follow a pulmonary rehabilitation program afterwards.

Main study parameters: The main study parameter is the difference in change in endurance time measured by an endurance cycle test between the EBV treatment group and the bronchoscopic lung volume reduction + rehabilitation group (EBV+PR).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: This study has no major risks for the participating patients. The patients will be exposed to additional exercise capacity and physical activity measurements, 3 additional questionnaires, a CT scan of the quadriceps muscle, a DEXA scan and peripheral blood collection. Furthermore, a subgroup of patients will be exposed to a cardiac MRI or muscle and fat biopsies. Patient can directly benefit from the EBV treatment and the pulmonary rehabilitation program. Indirect benefit might be achieved, because, at a group level the investigators will learn more about this novel treatment for our severe emphysema patients and will be able to further optimize this treatment.

ELIGIBILITY:
Inclusion Criteria:

* COPD.
* FEV1 ≤45%pred AND FEV1/FVC <70%.
* TLC >100%pred AND RV>175%pred.
* CAT ≥18.
* >50% emphysema destruction @-910HU.
* >95% complete major fissure measured by quantitative CT analysis.
* Non-smoking >6 months.
* Signed informed consent.

Exclusion Criteria:

* PaCO2>8.0 kPa, or PaO2<6.0kPa.
* 6-minute walk test <160m.
* Significant chronic bronchitis, bronchiectasis, or other infectious lung disease.
* 3 of more hospitalizations due to pulmonary infection within last 12 months before baseline assessments
* Previous lobectomy, LVRS, or lung transplantation.
* LVEF<45% and or RVSP>50mmHg.
* Anticoagulant therapy which cannot be weaned off prior to procedure.
* Patient is significantly immunodeficient.
* Involved in other pulmonary drug studies within 30 days prior to this study.
* Pulmonary nodule which requires intervention
* Any disease or condition that interferes with completion of initial or follow-up assessments

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Endurance time | After 6 months
  The difference in change in endurance time measured by an endurance cycle test between the EBV treatment group and the bronchoscopic lung volume reduction + rehabilitation group (EBV+PR).

SECONDARY OUTCOMES:
Pulmonary rehabilitation1 | After 6 months
  • the difference between the EBV treatment group and the EBV+PR group in change in:
  * Physical activity measured by accelerometry
Pulmonary rehabilitation2 | After 6 months
  • the difference between the EBV treatment group and the EBV+PR group in change in:
  * Lung function measured by bodyplehtysmography
Pulmonary rehabilitation3 | After 6 months
  • the difference between the EBV treatment group and the EBV+PR group in change in:
  * Exercise capacity measured by an 6-minute walk distance test
Patient reported outcomes | After 6 months
  • the change after EBV treatment in fatigue level measured by the CIS questionnaire.
Cardiopulmonary function | After 8 weeks
  • the change after EBV treatment in RVEDVI as measured with cardiac MRI.
Metabolism and change in body composition | After 8 weeks
  • the change after EBV treatment in fat-free mass index, fat mass, and fat distribution measured by a dexa scan.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk-Jan Slebos, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (2):
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - CIRO, Horn

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Posthuma R, van der Molen MC, Vaes AW, Hartman JE, Spruit MA, Slebos DJ, Vanfleteren LEGW. The impact of bronchoscopic lung volume reduction with endobronchial valves with or without pulmonary rehabilitation on symptoms of fatigue, anxiety and depression: a multicentre randomised controlled trial. ERJ Open Res. 2025 Aug 11;11(4):00892-2024. doi: 10.1183/23120541.00892-2024. eCollection 2025 Jul. PMID 40791921
- [Derived] van der Molen MC, Hartman JE, Vanfleteren LEGW, Kerstjens HAM, van Melle JP, Willems TP, Slebos DJ. Reduction of Lung Hyperinflation Improves Cardiac Preload, Contractility, and Output in Emphysema: A Clinical Trial in Patients Who Received Endobronchial Valves. Am J Respir Crit Care Med. 2022 Sep 15;206(6):704-711. doi: 10.1164/rccm.202201-0214OC. PMID 35584341